CLINICAL TRIAL: NCT01716286
Title: Neural Correlates of an Olive Oil Essence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Research Foundation (Other); German Federation of Industrial Research Associations (Other); Zentrum für Ernährungsmedizin und Prävention (Other); German Center for Diabetes Research (Other); University of Hohenheim (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Sabine Frank, Principal Investigator, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: YOG2
Record Dates: First submitted 2012-10-18; First posted 2012-10-29 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Neural Correlated of Different Foods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- yoghurt type (Experimental): low fat yoghurt vs. essence yoghurt
  Interventions: Dietary Supplement: low fat vs. essence yoghurt

INTERVENTIONS:
Dietary Supplement: low fat vs. essence yoghurt

SUMMARY:
The aim of the current study was to investigate the effect of a low fat meal in comparison to a low fat meal dosed with the fatfree essence of olive oil.

ELIGIBILITY:
Inclusion Criteria:

* male
* heatly

Exclusion Criteria:

* lactose intolerance
* fMRI cotraindications

Ages: 20 Years to 33 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
change in brain activity (cerebral blood flow change after yogurt intake) | 30 minutes before as well as 30 minutes and 120 minutes after yoghurt intake

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Tuebingen, MEG Center, Tübingen, Germany

REFERENCES:
- [Derived] Frank S, Linder K, Fritsche L, Hege MA, Kullmann S, Krzeminski A, Fritsche A, Schieberle P, Somoza V, Hinrichs J, Veit R, Preissl H. Olive oil aroma extract modulates cerebral blood flow in gustatory brain areas in humans. Am J Clin Nutr. 2013 Nov;98(5):1360-6. doi: 10.3945/ajcn.113.062679. Epub 2013 Sep 11. PMID 24025630